CLINICAL TRIAL: NCT07062315
Title: Impact of Chronotype-Based Time-Restricted Eating on Visceral Fat and Metabolic Health in Physically Inactive Adults With Central Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dai Zihan, Principal investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTEC-2025-189
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Central Obesity; Time Restricted Eating
MeSH Terms: conditions — Obesity, Abdominal; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chronotype-matched TRE (Experimental): Participants will eat ad libitum within an 8-hour eating window that match their chronotype.
  Interventions: Behavioral: Chronotype-matched time-restricted eating
- Chronotype-unmatched TRE (Active Comparator): Participants will eat ad libitum within an 8-hour eating window that unmatch their chronotype.
  Interventions: Behavioral: Chronotype-unmatched time-restricted eating
- Waitlist control (No Intervention): Participants in the waitlist control group will be instructed to maintain their previous eating or physical activity habits during the 12-week intervention. They will not receive any specific dietary advice or guidance. Weekly check-ins will be conducted to confirm continued participation and adherence. If they wish to participate, we will provide a suitable intervention after the duration of the study period.

INTERVENTIONS:
Behavioral: Chronotype-matched time-restricted eating — A 12 weeks time-restricted eating intervention that match participants' chronotype
  Arms: Chronotype-matched TRE
Behavioral: Chronotype-unmatched time-restricted eating — A 12 weeks time-restricted eating intervention that not match participants' chronotype
  Arms: Chronotype-unmatched TRE

SUMMARY:
Time-restricted eating (TRE) has gained attention as a promising dietary strategy for enhancing body composition and metabolic health. This innovative eating pattern involves confining daily food intake to a specific window, typically spanning 6-10 hours. Given the lack of consensus on the optimal TRE strategy, this research explores whether tailoring eating windows to individual chronotypes enhances TRE outcomes. This randomized controlled trial aims to evaluate the effects of chronotype-matched versus chronotype-unmatched TRE protocols, compared to a control group, over a 12-week period on visceral fat mass and other metabolic health outcomes in physically inactive adults with central obesity. Additionally, the study seeks to determine whether chronotype-matched TRE offers greater benefits in terms of visceral fat reduction and metabolic improvements compared to chronotype-unmatched TRE. Assessments will be conducted at baseline, and after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults, male or female, aged between 18-65 years old;
2. BMI of 23 kg/m² or higher, with a waist circumference exceeding 80 cm for females and 90 cm for males;
3. Weight stability for at least three months prior to the start of the study;
4. Physically inactive, indicated by not meeting established WHO guidelines on physical activity and sedentary behavior (i.e., at least 150-300 minutes of moderate-intensity or at least 75-150 minutes of vigorous-intensity aerobic exercise; or an equivalent combination of moderate and vigorous-intensity activity throughout the week;
5. Baseline eating duration exceeding 12 hours per day;
6. Identified as either early or late chronotypes (Morningness-Eveningness Questionnaire)

Exclusion Criteria:

1. Individuals currently or chronically receiving pharmacological treatment for hypertension, diabetes, weight loss, or other metabolic conditions;
2. Night shift workers;
3. Individuals with eating disorders;
4. Female participants who are breast-feeding, pregnant, or attempting to become pregnant;
5. Individuals currently participating in other weight-management programs or following other prescribed diet programs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Visceral fat mass | 12 weeks
  Visceral fat mass will be assessed using Magnetic Resonance Imaging (MRI)

SECONDARY OUTCOMES:
Subcutaneous fat mass | 12 weeks
  Subcutaneous fat mass will be assessed using Magnetic Resonance Imaging (MRI)
Body weight | 12 weeks
  Body weight (kg) will be measured by a bioelectrical impedance analyzer (BIA) with minimum clothing.
Body mass index (BMI) | 12 weeks
  BMI (kg/m2) will be calculated using body weight (kg) and height (m)
Body composition (Fat mass, fat free mass) | 12 weeks
  Body composition including fat mass and fat-free mass (kg) will be measured by bioelectrical impedance analyzer (BIA) with minimum clothing.
Anthropometric measures | 12 weeks
  Waist and hip circumferences (cm) will be assessed by standard procedures using a tension tape accurate to 0.1 cm. The waist-hip ratio will be calculated accordingly.
Fasting glucose metabolism | 12 weeks
  Fasting blood samples will be used to analyze biomarkers of glucose metabolism, including fasting glucose (mmol/L), fasting insulin (mU/L), HbA1c (mmol/mol), as well as derived indices (HOMA-IR) calculated from fasting glucose and insulin levels.
Fasting lipid metabolism | 12 weeks
  Fasting blood samples will be used to analyze different biomarkers of lipid metabolism including triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol (mmol/L)
Dietary patterns | 12 weeks
  Dietary pattern including eating window and dietary intake will be assessed using a seven-day food record
Subjective sleep quality | 12 weeks
  Subjective sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI)
Objectively sleep quality | 12 weeks
  Objectively sleep quality will be assessed by accelerometer
Subjective quality of life | 12 weeks
  Quality of life will be assessed through questionnaires (WHOQOL-BREF)
Appetite | 12 weeks
  Appetite will be measured by visual analog scale (VAS).

OTHER OUTCOMES:
Objectively physical activity levels | 12 weeks
  Objectively physical activity levels will be assessed by accelerometer, including time spent in sedentary behavior and moderate-to-vigorous physical activity (MVPA).
Chronotype | 12 weeks
  Chronotype will be assessed through Morningness-Eveningness Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Science and Physical Education, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No